CLINICAL TRIAL: NCT06097767
Title: Evaluation of the Incidence of Necrotizing Enterocolitis in Preterm Infants With Respiratory Distress Syndrome Undergoing Caffeine Therapy
Brief Title: the Incidence of Necrotizing Enterocolitis in Preterm With Respiratory Distress Syndrome Undergoing Caffeine Therapy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Gellan Alaa Mohamed Kamel Morsy, Lecturer of pharmacology and toxicology, Al-Azhar University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHDIRB2018122001/2116
Record Dates: First submitted 2023-10-13; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Pharmacological Action of Drug
MeSH Terms: interventions — caffeine citrate; Amikacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (Other): It includes preterm infants with respiratory distress syndrome aged 32 weeks-35 weeks receives regular intervention for RDS
  Interventions: Drug: Amikacin
- Caffeine-treated group (Active Comparator): It includes preterm infants with respiratory distress syndrome who received caffeine treatment as intravenous caffeinospire (Caffeine citrate) 60 mg / 3 ml (20 mg /ml) 3 ml vial for injection.
  Interventions: Drug: Caffeine citrate

INTERVENTIONS:
Drug: Caffeine citrate — It includes preterm infants with respiratory distress syndrome who received caffeine treatment as intravenous caffeinospire (Caffeine citrate) 60 mg / 3 ml (20 mg /ml) 3 ml vial for injection.
  Arms: Caffeine-treated group
Drug: Amikacin — it includes preterm infants with respiratory distress syndrome who received amikacin in regular intervention therapy in control group
  Arms: Control group

SUMMARY:
It is a randomized, prospective study; it will be carried out in the NICU at Alzahraa University Hospital including 50 newborn babies diagnosed with respiratory distress syndrome.

The purpose of this study is to :

1. Investigate the protective caffeine on necrotizing enterocolitis in respiratory distress syndrome preterm infants.
2. Detect the impact of caffeine protocol treatment on the in-incidence of necrotizing enterocolitis in respiratory distress syndrome preterm infants in neonatal intensive care

1- Control group It includes preterm infants with respiratory distress syndrome aged 32 weeks-35 weeks.

2- Caffeine-treated group It includes preterm infants with respiratory distress syndrome who received caffeine treatment as intravenous caffeinospire (Caffeine citrate) 60 mg / 3 ml (20 mg /ml) 3 ml vial for injection.

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants with respiratory distress syndrome.

Exclusion Criteria:

* Preterm admitted to NICU for other reasons rather than respiratory distress
* Major congenital anomalies
* spontaneous intestinal perforation
* Endocrinal Dysfunctions

Ages: 32 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
decreasing NEC rates | 1 year
  decreasing NEC rates and stage ≥2 and death.

CONTACTS AND LOCATIONS:
Locations (1):
- NICU at Alzahraa University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided